CLINICAL TRIAL: NCT00963365
Title: Pt. A: Ph I, Sngl-Blind, Randomized, Pcbo-Controlled 3-Way Crossover Study Followed by an Open-label Food Effect Study to Assess the PK of IV and Oral AZD6765 in Healthy Male and Female Subjects Pt.B: Ph I, Double-Blind, Randomized, Placebo-Controlled Study to Assess the Safety, Tolerability and PK of AZD6765 When Administered in Multiple Ascending Doses to Healthy Subjects
Brief Title: AZD6765 Oral Single Ascending Dose/Multiple Ascending Dose (SAD/MAD)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: D6703C00001
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Phase 1; Healthy volunteers
MeSH Terms: interventions — AZD6765

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- AZD6765 oral solution (Experimental): Active
  Interventions: Drug: AZD6765
- AZD6765 IV infusion (Experimental): Active
  Interventions: Drug: AZD6765
- Placebo to AZD6765 oral solution (Placebo Comparator): Placebo
  Interventions: Drug: AZD6765
- Placebo to AZD6765 IV infusion (Placebo Comparator): Placebo
  Interventions: Drug: AZD6765

INTERVENTIONS:
Drug: AZD6765 — Single oral dose and single IV infusion of AZD6765
Drug: AZD6765 — Once-daily oral dose of AZD6765 or placebo on Day 1 and on Days 4 through 9.
  Arms: AZD6765 oral solution; Placebo to AZD6765 oral solution

SUMMARY:
The purpose of this study is to determine the safety of AZD6765 when given in single and multiple oral doses and to compare an oral and intravenous (IV) formulation of AZD6765 to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Females must be of non-childbearing potential.

Exclusion Criteria:

* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational product.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment within 3 months (if half-life was < 24 hours) of the first administration of study drug
* Plasma or blood product donation within one month of screening or any blood donation/blood loss > 500mL during the 3 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
The objective of the study is to investigate the safety and tolerability of AZD6765 when administered orally in single and multiple doses to healthy subjects by assessment of adverse events, vital signs, physical examinations, electrocardiograms(ECG). | Safety assessments are made prior to and after drug administration.

SECONDARY OUTCOMES:
Part A 1. To characterize the single dose pharmacokinetics of AZD67652. To assess the absolute bioavailability of AZD67653. To assess the effect of food on the pharmacokinetics of AZD6765 | Blood samples will be obtained on Days 1-5.
Part B 1. To characterize the single and multiple dose pharmacokinetics of AZD6765 2. To assess dose linearity and proportionality of AZD67653. To assess the degree of accumulation and the time dependence of the pharmacokinetics of AZD6765 | Blood samples will be obtained on Days 1-4 and 7-11.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Leese, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, Overland Park, Kansas, United States